CLINICAL TRIAL: NCT05238948
Title: A Phase 1, Open-label, 1-sequence Crossover Drug-drug-interaction Study to Assess the Effect of Single and Multiple Doses of CKD-506 on the Single-Dose Pharmacokinetics of Midazolam, A CYP3A4 Substrate, in Healthy Male Subjects
Brief Title: CKD-506 Drug-Drug Interaction Study in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: A82_04DDI2124; 2021-006496-41 (EudraCT Number)
Record Dates: First submitted 2022-01-11; First posted 2022-02-14 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-01

CONDITIONS: Drug Drug Interaction
Keywords: CYP3A4; Midazolam
MeSH Terms: interventions — Midazolam; CKD-506; Single Person

STUDY DESIGN:
Intervention Model Description: One arm and 1-sequence crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Midazolam with/without CKD-506 (Experimental): Single arm and 1-sequence crossover
  Interventions: Drug: Midazolam; Drug: CKD-506

INTERVENTIONS:
Drug: Midazolam — Substrate of CYP3A4
  Other Names: Single dose
Drug: CKD-506 — Perpetrator of CYP3A4
  Other Names: Single and multiple dose

SUMMARY:
This will be a Phase 1, open-label, 1-sequence crossover drug-drug-interaction study in 16 healthy male subjects to assess the effect of single and multiple doses of CKD-506 on the single-dose PK of oral midazolam. Midazolam will be used as a cytochrome P450 (CYP)3A4 substrate in this study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects
* Ability and willingness to abstain from methylxanthine-containing beverages or food (coffee, tea, cola, chocolate, energy drinks)
* Ability and willingness to abstain from foods and beverages containing grapefruit, Seville oranges, pomelos, star fruit, or cranberries

Exclusion Criteria:

* History of relevant drug and/or food allergies.
* Using tobacco products
* Positive drug and alcohol screen

Ages: 20 Years to 49 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only male subjects are eligible.
Enrollment: 17 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-04-29 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of oral midazolam | For 24 hours
  With and without coadministration of CKD-506
Area Under Curve (AUC) of oral midazolam | For 24 hours
  With and without coadministration of CKD-506

SECONDARY OUTCOMES:
Cmax of CKD-506 and its metabolites following oral single and multiple doses of CKD-506 | For 24 hours
AUC of CKD-506 and its metabolites following oral single and multiple doses of CKD-506 | For 24 hours
Time to Maximum Plasma Concentration (Tmax) of CKD-506 and its metabolites following oral single and multiple doses of CKD-506 | For 24 hours
Number of treatment emergent adverse events | Over 4 weeks
  assessed by clinical laboratory, vital signs, 12-lead electrocardiogram, and physical examination
Number of participants with treatment emergent adverse events | Over 4 weeks
  assessed by clinical laboratory, vital signs, 12-lead electrocardiogram, and physical examination

CONTACTS AND LOCATIONS:
Overall Officials: Maria Velinova,, MD, PhD, Principal Investigator — PRA Group BV, a PRA Health Sciences company
Locations (1):
- PRA Health Sciences, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No